CLINICAL TRIAL: NCT06852404
Title: Understanding Death: The Impact of Cultural Factors on Nursing Students' Perception of Death
Brief Title: Understanding Death: Cultural Factors Affecting Nursing Students' Perception
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nursemin ÜNAL, Associate Professor, Ankara University
Other Study IDs: 2025
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Nursing Education; Death; Cultural Factors
Keywords: cultural factors; transcultural care; death; nursing students
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Photovoice — Photovoice is a participant-driven research method that enables individuals to communicate their experiences through visual data. It is especially useful for exploring social issues and the challenges people encounter. In this approach, participants capture images that they find meaningful in relation to the research topic, using these photographs to express their emotions, thoughts, and personal experiences.

SUMMARY:
Cultural factors play a key role in shaping individuals' perceptions of death, alongside personal beliefs, professional experience, and education. Nursing students must balance their personal and cultural values with their professional responsibilities, as cultural differences influence attitudes toward death and mourning. Understanding nursing students' perceptions of death is crucial for enhancing their education and professional competence. Integrating cultural perspectives into nursing education can help students develop a more conscious and prepared approach to end-of-life care. This study aims to explore the impact of cultural factors on nursing students' perceptions of death and propose strategies to enhance cultural sensitivity in education.

DETAILED DESCRIPTION:
Death is a universal phenomenon with varying meanings at both individual and societal levels. Today, most deaths occur in hospitals, highlighting the critical role of nurses in end-of-life care. However, research indicates that patient death is a significant source of stress for nursing students, who often feel unprepared to cope with it. Cultural factors play a key role in shaping individuals' perceptions of death, alongside personal beliefs, professional experience, and education. Nursing students must balance their personal and cultural values with their professional responsibilities, as cultural differences influence attitudes toward death and mourning. Some cultures openly discuss death, while others consider it a taboo, affecting students' experiences and emotional responses. Understanding nursing students' perceptions of death is crucial for enhancing their education and professional competence. Integrating cultural perspectives into nursing education can help students develop a more conscious and prepared approach to end-of-life care.

This study aims to explore the impact of cultural factors on nursing students' perceptions of death and propose strategies to enhance cultural sensitivity in education. Using the photo storytelling method, it will examine how students shape their perceptions of death through visual and narrative expressions, fostering deeper cultural awareness and emotional resilience in their professional practice. In this study, students meeting the inclusion criteria will be informed about the research's purpose and method and invited to participate. Those who agree will complete a Demographic Information Form. Participants will then be asked to submit three self-taken photos reflecting their perception of death within one week. Before taking the photos, they will receive guidelines on the procedure. Photos, along with date, time, and brief descriptions, will be sent via email to the lead researcher. The collected photos will be securely stored on the researcher's personal computer, coded, and preserved with transcripts for use during interviews.

ELIGIBILITY:
Inclusion Criteria:

* Be a third-year student in the Nursing Department of a Health Sciences Faculty at a university in Ankara during the 2024-2025 academic year
* Own a smartphone capable of taking photographs
* Be willing to participate in the study.

Exclusion Criteria:

* Students who wish to withdraw from the study at any stage will not be included in the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of third-year students enrolled in the Nursing Department program at a private university.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Semi-structured Questions | Within 1 week after participating in the study and submitting the photos to the researcher]
  This semi-structured interview explores personal and cultural perceptions of death, reflections on participant-taken photos, and the impact of these experiences on nursing students' views and professional readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Nursemin Unal, Assoc. Prof., Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng R, Guo Q, Dong F, Gao L. Death Self-efficacy, Attitudes Toward Death and Burnout Among Oncology Nurses: A Multicenter Cross-sectional Study. Cancer Nurs. 2022 Mar-Apr 01;45(2):E388-E396. doi: 10.1097/NCC.0000000000000839. PMID 32511153
- [Background] Petrongolo M, Toothaker R. Nursing students perceptions of death and dying: A descriptive quantitative study. Nurse Educ Today. 2021 Sep;104:104993. doi: 10.1016/j.nedt.2021.104993. Epub 2021 May 28. PMID 34098421
- [Background] Wang C, Burris MA. Photovoice: concept, methodology, and use for participatory needs assessment. Health Educ Behav. 1997 Jun;24(3):369-87. doi: 10.1177/109019819702400309. PMID 9158980
- [Background] Randall PS, De Gagne JC, Yamane SS, Lee E. The use of photovoice in nursing education: A scoping review. Nurs Health Sci. 2023 Dec;25(4):516-529. doi: 10.1111/nhs.13057. Epub 2023 Oct 14. PMID 37837266
- [Background] Wang Y, Jin X, Liu M. Nursing students' perceptions of a good death: A mixed method study. Nurse Educ Today. 2024 Nov;142:106343. doi: 10.1016/j.nedt.2024.106343. Epub 2024 Aug 5. PMID 39126999